CLINICAL TRIAL: NCT01181622
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, 7-Day Safety and Tolerability Study of Denufosol Tetrasodium Inhalation Solution Administered Via PARI LC® Star in Patients 2 to 4 Years of Age With Cystic Fibrosis
Brief Title: A Safety and Tolerability Study of Denufosol in 2-4 Year Olds
Acronym: REACH-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P08643; 08-116
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- denufosol tetrasodium Inhalation Solution (Experimental)
  Interventions: Drug: denufosol tetrasodium Inhalation Solution
- Placebo (Placebo Comparator)
  Interventions: Drug: 0.9% w/v sodium chloride solution

INTERVENTIONS:
Drug: denufosol tetrasodium Inhalation Solution — 60 mg by oral inhalation three times daily
  Arms: denufosol tetrasodium Inhalation Solution
Drug: 0.9% w/v sodium chloride solution — 0.9% w/v sodium chloride solution by oral inhalation three times daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of denufosol 60 mg TID in pediatric CF patients 2 to 4 years of age

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of CF
* Have oxyhemoglobin saturation ≥ 95% prior to randomization

Exclusion Criteria:

* Have acute intercurrent respiratory infection (cough, wheezing, or new

rhinorrhea or nasal congestion)

* Have any significant medical condition not related to CF
* Unable to discontinue use of hypertonic saline

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Intolerability to study drug as measured by: oxyhemoglobin saturation, treatment-emergent cough, and new wheezes or crackles | Day 1, Day 7

SECONDARY OUTCOMES:
Mean change from pre-dose in oxyhemoglobin saturation at defined times post-dose | Day 1, Day 7
Mean change from baseline in oxyhemoglobin saturation | Day 7
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs) and/or withdrawals due to TEAEs | Day 7
Mean change from pre-dose in pulse and respiratory rate at defined times post-dose | Day 1, Day 7
Mean change from baseline in pulse and respiratory rate | Day 7
Incidence of new medical condition(s) or worsening of previous medical condition(s) from baseline | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Smiley, MD, Study Director — Medical monitor